CLINICAL TRIAL: NCT06287541
Title: A Prospective, Multicenter, Randomized Study Comparing the Necessity of a Second Transurethral Resection of Bladder Tumor in High-risk Non-muscle-invasive Bladder Cancer Patients With Negative Urine Biomarker After Initial Transurethral Resection
Brief Title: The Necessity of a Second Transurethral Resection in High-risk Non-muscle-invasive Bladder Cancer Patients With Negative Urine Biomarker After Initial Transurethral Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Qiang Lv, Principal Investigator, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SR-486
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Non Muscle Invasive Bladder Cancer
Keywords: reTURBT; NMIBC; urine biomarker; RFS
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Fanconi Syndrome

STUDY DESIGN:
Intervention Model Description: Participants who meet the inclusion criteria are randomized 1:2 into two parallel groups. Group A: Participants assigned to this group will not undergo reTURBT. They will receive standard follow-up care as per institutional guidelines.
  Group B: Participants assigned to this group will undergo reTURBT as part of their treatment protocol. Following reTURBT, they will also receive standard follow-up care. Outcome measures of recurrence rate and RFS would be compared between the two groups to determine the effectiveness and safety of the urine genetic test-guided approach compared to standard care with reTURBT.Throughout the study period, both groups are followed up simultaneously, allowing for parallel comparisons of outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urine biomarker -Guided without reTURBT (Experimental): Participants in this arm will proceed without reTURBT.
  Interventions: Procedure: Urine biomarker -Guided without reTURBT
- Standard Care with reTURBT (No Intervention): Participants in this arm will receive standard care, which undergo reTURBT

INTERVENTIONS:
Procedure: Urine biomarker -Guided without reTURBT — Participants will proceed without reTURBT
  Arms: Urine biomarker -Guided without reTURBT

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of using a urine biomarker test to guide the decision-making process regarding the necessity of reTURBT in NMIBC patients. The main question aims to answer whether patients with negative urine biomarker tests can safely avoid reTURBT without compromising recurrence-free survival. Participants who have completed the initial TURBT and tested negative for the urine biomarker will be enrolled in the study. They will then be randomized 1:2 into two groups:Group A: Participants will not receive reTURBT and Group B: Participants will undergo reTURBT. Researchers will compare the RFS rates between Group A (no reTURBT) and Group B (reTURBT) to determine if the urine biomarker test can safely spare patients from unnecessary reTURBT.

DETAILED DESCRIPTION:
This clinical trial aims to address the clinical question of whether a urine biomarker test can effectively guide the decision-making process regarding the necessity of reTURBT (repeat transurethral resection of bladder tumor) in patients with non-muscle-invasive bladder cancer (NMIBC). The primary objective is to assess whether patients with negative urine biomarker tests can safely avoid reTURBT. Participants eligible for enrollment in this study will be randomized in a 1:2 ratio into two groups:Group A: Participants assigned to this group will not undergo reTURBT. They will receive standard follow-up care as per institutional guidelines. Group B: Participants assigned to this group will undergo reTURBT. Following reTURBT, they will also receive standard follow-up care. The main task for participants will involve providing urine samples for the biomarker test before reTURBT. Those in Group B will additionally undergo reTURBT, a standard surgical procedure involving the removal of residual tumor tissue from the bladder.Throughout the study period, researchers will assess their recurrence-free survival rates and RFS. The goal is to determine whether the urine biomarker test can safely spare patients from unnecessary reTURBT while maintaining comparable RFS rates. This study adheres to ethical guidelines and has obtained approval from the appropriate institutional review boards. Participant confidentiality and data integrity will be strictly maintained throughout the study duration. The results of this trial have the potential to inform clinical practice guidelines and improve the management of NMIBC patients by offering a personalized approach to treatment decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NMIBC who have undergone initial TURBT and are scheduled for reTURBT surgery as recommended by guidelines or chosen by their physicians;
* Patients who have tested negative for urine biomarkers after the initial TURBT and before the second TURBT;
* Age ≥ 18 years;
* Willingness to provide personal basic clinical information, as well as pathology and subsequent recurrence monitoring results;
* Willingness to sign informed consent.

Exclusion Criteria:

* Patients with other non-urothelial malignant tumors (including prostate cancer and renal cell carcinoma);
* Patients previously diagnosed with muscle-invasive bladder cancer;
* Patients unable to undergo a second transurethral resection;
* Patients with incomplete sample pathology information;
* Any condition perceived by the researcher to potentially harm the subjects or prevent them from meeting or executing the study requirements;
* Patients unable to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
2-year RFS rate | from initial TURBT to the first confirmed recurrence within 2 years
  the proportion of participants experiencing a recurrence during follow-up within 2 years

SECONDARY OUTCOMES:
RFS | from initial TURBT to the first confirmed recurrence within 2 years
  the duration from the completion of initial TURBT until the first recurrence of cancer is detected or until the end of the follow-up period, whichever comes first.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR
Time Frame: by 2029 for 5 years
Access Criteria: will be shared under request
URL: https://www.ncbi.nlm.nih.gov